CLINICAL TRIAL: NCT00950846
Title: Umbilical Cord Blood Transplant for Congenital Pediatric Disorders
Acronym: UCB
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Baylor College of Medicine (Other)
Collaborators: Center for Cell and Gene Therapy, Baylor College of Medicine (Other)
Responsible Party: Principal Investigator, Caridad Martinez, Assistant Professor, Pediatric Hematology/Oncology, Center for Cell and Gene Therapy, Baylor College of Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25064-UCB
Record Dates: First submitted 2009-07-30; First posted 2009-08-03 (Estimated); Results first posted 2023-10-30 (Actual); Last update posted 2023-10-30 (Actual); Status verified 2023-10

CONDITIONS: Congenital Pediatric Disorders
Keywords: Congenital Pediatric Disorders; Umbilical Cord Blood Transplant; Congenital Abnormalities; Cord Blood Stem Cell Transplantation; Busulfan; Cytoxan; Cyclophosphamide; Fludarabine
MeSH Terms: conditions — Congenital Abnormalities | interventions — Busulfan; Cyclophosphamide; fludarabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Umbilical Cord Blood Transplant Treatment Plan (Experimental): Busulfan, Cytoxan, Fludarabine, Cord Blood Stem Cell Infusion
  Interventions: Drug: Busulfan; Drug: Cytoxan; Drug: Fludarabine; Procedure: Cord Blood Stem Cell Infusion

INTERVENTIONS:
Drug: Busulfan — Day -9, -8, -7 and -6
  Patients less than or equal to 12 kg: 1.1 mg/kg/dose IV every 6 hours for 16 doses total; patients >12 kg: 0.8 mg/kg/dose IV every 6 hours for 16 doses.
  Other Names: Busulfex
Drug: Cytoxan — (50 mg/kg/dose) will be given IV on Days -5, - 4, -3, and -2 over 2 hours (can be given over 1 to 4 hours as determined by the treating physician). The total dose to be given over 4 days is 200 mg/kg.
  Other Names: Cyclophosphamide
Drug: Fludarabine — 40 mg/m2/day IV over 1 hour for patients greater than 10 kg, or 1.3 mg/kg/day for patients less than or equal to 10 kg.
  Other Names: Fludera
Procedure: Cord Blood Stem Cell Infusion — The cord blood stem cells will be infused on Day 0.

SUMMARY:
The purpose of this study is to determine the safety and effectiveness of Umbilical Cord Blood Transplant (UCBT) to treat the patient's disease, and to see if this treatment can decrease the incidence of GVHD.

This study is for patients that were born with a disease that affects their body's metabolism or immune system. The doctor plans to treat the patient for this illness with a stem cell transplant.

While improved medical care has allowed many people with these diseases to live longer, the only way to truly cure the diseases is by means of a stem cell transplant from a donor who does not have the disease. A stem cell transplant will replace sick cells with new healthy donor cells. Stem cells grow into different types of blood cells that people need, including red blood cells, white blood cells, and platelets. In a stem cell transplant, the patients own stem cells would be killed by chemotherapy drug and then replaced by stem cells from the donor. Stem cells can be collected from the bone marrow, peripheral blood or umbilical cords. In this study, umbilical cords will be the source of the stem cells.

Currently, large inventories of umbilical cord blood units are available in public banks for transplantation in those lacking bone marrow donors. UCB transplants offer several advantages over adult bone marrow or peripheral blood stem cell transplants, including:

1. Rapid availability,
2. Absence of donor risk,
3. Low risk of transmissible infectious diseases,
4. Low risk of acute GvHD (as compared to recipients of unrelated donor marrow and peripheral blood cells).

The two main causes of death after umbilical cord blood transplantation for disorders for these kinds of patients, are graft failure and infection.

In this study we are trying to address these two problems by using different drugs to prepare patients for the transplant.

To help improve engraftment (cells begin to grow), we will include the drug Fludarabine to the usually used Busulfan and Cytoxan that the study patients will receive before their transplant.

We will try to decrease the chance of developing graft-versus-host disease (GvHD) by using Cyclosporin A (CSA) and Mycophenolate Mofetil (MMF), instead of Anti-Thymocyte Globulin (ATG) which is normally used.

DETAILED DESCRIPTION:
Patients will be examined to make sure that they meet the requirements of this study. There will be tests of the heart and of the lungs. X-rays will be taken of the lungs and other organs, depending on the disease. An MRI and consultations with different specialists will also be conducted.

Patients also must have a negative pregnancy test before entering this study if they are a woman of childbearing potential. The blood will be tested for viruses and to look at the functioning of the liver and kidneys. The examination also includes HIV testing. If the patient has HIV, they will not be able to be treated on this protocol.

After we have determined that the patient is eligible for treatment on this study and a suitable UCB stem donor has been found, they will have a central line placed.

After placement of the central line, the following chemotherapy will be given to after admission to the hospital:

* 9 days before the infusion through 6 days before the infusion: Busulfan every 6 hours for 16 total doses.
* 5 days before the infusion through 2 days before the infusion: Cytoxan given daily for 4 days over 2 hours. (It can be given over 1 to 4 hours if needed as decided by the physician). Mesna will be given per standards.
* 4 days before the infusion through 1 day before the infusion: Fludarabine given daily for 4 days over 1 hour.

Stem cell transplant (infusion of the UCB stem cells) - defined as Day 0 of the treatment. All other "numbered" days relate to this infusion date. For example, Day 1 is the first day after the stem cell transplant.

Standard Therapy: Phenytoin will be given according to the standards of the TCH formulary.

Cyclosporin A (CSA) will be given starting 2 days prior to the stem cell infusion. It will be given daily over 2 hours every 12 hours, and then tapered if no GvHD is present.

Administration of Mycophenolate Mofetil (MMF) will start on the day the stem cell infusion is completed, and will continue daily for 45 days unless the patient develops GvHD.

Intravenous Immunoglobulins (IVIG) will be given as per CAGT SOP for infections prophylaxis.

Granulocyte Colony-Stimulating Factor (GCSF) will be given daily starting at Day +7 until ANC is greater than 2,500 for three consecutive days.

Study Evaluation: Patients will have various study evaluations, including blood samples, before and after the transplant.

Follow-Up: After year 1, the patients will be asked to return to the clinic once a year for consultations. These consultations with specialists will be similar to the ones the patients had before their transplant.

ELIGIBILITY:
INCLUSION CRITERIA:

* Patients less than 18 years of age.
* Patients with a congenital or acquired immunologic, hematological, or metabolic pediatric disease (including SCID) in which stem cell transplantation has been beneficial.
* Related or Unrelated Umbilical Cord Blood Unit with 0-1 antigen mismatch, 5-6 HLA- A and B (at low to intermediate resolution) and DRB1 (at high resolution).
* Total cryopreserved HSC graft cell dose must be 5 x 10^7 or greater nucleated cells per kilogram recipient body weight.
* Lansky/Karnofsky scores 60 or greater.
* Patient has DLCO > 50% predicted or FEV1 > 50%, if applicable.
* Written informed consent and/or signed assent line from patient, parent or guardian.

EXCLUSION CRITERIA:

* Patients with uncontrolled infections as assessed by the principal investigator only. For bacterial infections, patients must be receiving definitive therapy and have no signs of progressing infection for 72 hours prior to starting conditioning. For fungal infections patients must be receiving definitive systemic antifungal therapy and have no signs of progressing infection for 1 week prior to enrollment. Progressing infection is defined as hemodynamic instability attributable to sepsis or new symptoms, worsening physical signs or radiographic findings attributable to infection. Persisting fever without other signs or symptoms will not be interpreted as progressing infection.
* Severe renal disease (creatinine > 3X normal for age).
* Severe hepatic disease (direct bilirubin > 3 mg/dL or SGOT > 500).
* Patients with symptomatic cardiac failure unrelieved by medical therapy or evidence of significant cardiac dysfunction by echocardiogram (shortening fraction < 20%).
* HIV positive.

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 40 (Actual)
Dates: Start 2009-09 (Actual); Primary Completion 2020-07-21 (Actual); Study Completion 2021-02-04 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Caridad Martinez, MD, Principal Investigator — Baylor College of Medicine
Locations (1):
- Texas Children's Hospital, Houston, Texas, United States

REFERENCES:
- [Derived] Martinez C, Aguayo-Hiraldo P, Chaimowitz N, Forbes L, Rider N, Nicholas S, Seeborg F, Chinen J, Chinn I, Davis C, Roseblatt H, Noroski L, Omer B, John T, Yassine K, Naik S, Craddock J, Bhar S, Allen C, Ahmed N, Sasa G, Steffin D, Doherty E, George A, Salem B, Friend B, Hegde M, Brenner MK, Heslop HE, Leen A, Pena A, Wu M, Hanson IC, Krance RA. Cord blood transplantation for nonmalignant disorders: early functional immunity and high survival. Blood Adv. 2023 May 9;7(9):1823-1830. doi: 10.1182/bloodadvances.2022009038. PMID 36453638

RESULTS

PARTICIPANT FLOW:
Groups:
- Umbilical Cord Blood Transplant Treatment Plan: Busulfan, Cytoxan, Fludarabine, Cord Blood Stem Cell Infusion
  Busulfan: Day -9, -8, -7 and -6
  Patients less than or equal to 12 kg: 1.1 mg/kg/dose IV every 6 hours for 16 doses total; patients >12 kg: 0.8 mg/kg/dose IV every 6 hours for 16 doses.
  Cytoxan: (50 mg/kg/dose) will be given IV on Days -5, - 4, -3, and -2 over 2 hours (can be given over 1 to 4 hours as determined by the treating physician). The total dose to be given over 4 days is 200 mg/kg.
  Fludarabine: 40 mg/m2/day IV over 1 hour for patients greater than 10 kg, or 1.3 mg/kg/day for patients less than or equal to 10 kg.
  Cord Blood Stem Cell Infusion: The cord blood stem cells will be infused on Day 0.
Period: Overall Study
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Started | 40
Completed | 30
Not Completed | 10
Not completed — Death | 6
Not completed — Lost to Follow-up | 3
Not completed — Possible undiagnosed AML at study entry | 1

BASELINE CHARACTERISTICS:
Population: The analysis included 38 evaluable participants who completed conditioning and received transplant. Two participants who were enrolled but considered not evaluable for the study were excluded from the analysis. One participant died before receiving transplant. The other was diagnosed with aplastic anemia without signs of malignancy at the time of enrollment, but later showed signs of MDS and progressed to AML, which made the participant not evaluable for this study.
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 38
Age, Continuous [Median (Full Range); unit: months] — Population: This is age at transplant. One participant did not receive transplant.
  months | 5 [1 to 111]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 15
  Male | 23
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 20
  Not Hispanic or Latino | 18
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 2
  White | 35
  More than one race | 0
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Overall Survival at 100 Days After Umbilical Cord Blood Transplant in Pediatric Patients.
Description: To determine the overall survival rate at 100 days after umbilical cord blood transplant in pediatric patients with myeloid hematological malignancies.
Time Frame: 100 days
Population: The analysis included 38 evaluable participants who completed conditioning and received transplants. Two participants were excluded from the analysis. One participant died before receiving transplant and the other was diagnosed with aplastic anemia without signs of malignancy at the time of enrollment, but later showed signs of MDS and progressed to AML, which made the participant not evaluable for this study.
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 38
probability of overall survival | 0.947 [0.806 to 0.987]

2. Primary Outcome: Overall Survival at 1 Year After Umbilical Cord Blood Transplant in Pediatric Patients.
Description: To determine the overall survival rate at 1 year after umbilical cord blood transplant in pediatric patients with myeloid hematological malignancies.
Time Frame: 1 year
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 38
probability of overall survival | 0.868 [0.712 to 0.943]

3. Primary Outcome: Overall Survival at 3 Years After Umbilical Cord Blood Transplant in Pediatric Patients.
Description: To determine the overall survival rate at 3 years after umbilical cord blood transplant in pediatric patients with myeloid hematological malignancies.
Time Frame: 3 years
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: probability of overall survival
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 38
probability of overall survival | 0.868 [0.712 to 0.943]

4. Secondary Outcome: Number of Participants With Platelet Engraftment
Description: Achievement of untransfused platelet count > 20 x 10^9/L on three consecutive days
Time Frame: Day 42
Population: The analysis included 37 evaluable participants who completed conditioning, received transplants and were alive on day 42. Three participants were excluded from the analysis. One participant died before receiving transplant, one was not evaluable due to possible undiagnosed AML at study entry, and one died on day 31 after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 37
Participants
  Engrafted | 17
  Not engrafted | 20

5. Secondary Outcome: Incidence of Severe Grade III-IV Acute GvHD at Day 100.
Description: Number of participants with acute GVHD graded by the method of Przepiorka et al, which evaluates skin involvement, lower and upper GI, and liver function (bilirubin), each being graded in stages from 0 to 4, where 0 means no acute GVHD, and 4 is the highest stage of acute GVHD.
Time Frame: Day 100
Population: The analysis included all participants who received transplants and were evaluable for acute GVHD. One participant was not evaluable due to possible undiagnosed AML at study entry and all other participants who received transplants were evaluable for acute GVHD if he/she engrafted and either completed 100 days observation after transplant or experienced acute GVHD.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 36
Participants | 1

6. Secondary Outcome: Number of Participants With Chronic GvHD
Description: Number of participants with chronic GVHD graded by the method of Przepiorka et al, which evaluates skin, joints, oral, ocular, hepatic, esophagus, GI, respiratory, platelet, and musculoskeletal involvement, in stages from 0 to 3.
Time Frame: 1 year
Population: The analysis included all participants who received transplants and were evaluable for chronic GVHD. One participant was not evaluable due to possible undiagnosed AML at study entry and all other participants who received transplants were evaluable for chronic GVHD if he/she engrafted and survived or remained in the study for more than 101 days after transplant.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 35
Participants | 1

7. Secondary Outcome: Number of Participants With Donor Engraftment After Transplant.
Description: To evaluate donor engraftment at 100 days, 6 and 12 months after transplant.
Time Frame: 100 days, 6 months and 12 months
Population: The analysis included all participants who underwent transplant and were evaluable at the time of assessments. One participant was not evaluable due to possible undiagnosed AML at study entry.
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 36
Participants
  100 days | 36
  6 months: number analyzed (Participants) | 33
  6 months | 33
  12 months: number analyzed (Participants) | 33
  12 months | 33

8. Secondary Outcome: Number of Participants With Neutrophil Engraftment
Description: Achievement of absolute neutrophil count > 0.5 x 10^9/L on three consecutive days
Time Frame: Day 42
Population: as for outcome 4
Measure: Count of Participants; unit: Participants
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
Number analyzed (Participants) | 37
Participants
  Engrafted | 37
  Not engrafted | 0

ADVERSE EVENTS:
Time Frame: We have recorded all grade 3 and 4 toxicities, except hematological toxicities, fever, abnormal glucose, ALT, GGT, and K levels from the day conditioning started until day 30 post-transplant. SAEs were reported up to day 100. Our study primary outcome is Overall Survival (OS) up to 3 years after transplant. The use of AEs up to 100 days is the standard measurement after a stem cell transplant. OS will capture any major toxicity up to 3 years after transplant that will lead to mortality.
Arm/Group | Umbilical Cord Blood Transplant Treatment Plan
All-Cause Mortality (participants affected / at risk) | 6/40
Serious Adverse Events (participants affected / at risk) | 27/40
Other Adverse Events (participants affected / at risk) | 25/40
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood Transplant Treatment Plan (N=40)
Acute kidney injury (Renal and urinary disorders) | 2 (2)
Blood and lymphatic system disorders - Other, specify: Thrombotic microangiopathy (Blood and lymphatic system disorders) | 1 (1)
Cardiac General - Other: Cardiopulmonary collapse of unknown etiology (Cardiac disorders) | 1 (1)
Cardiac arrest (Infections and infestations) | 1 (1)
Catheter related infection (Metabolism and nutrition disorders) | 8 (8)
Dehydration (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Dyspnea (Gastrointestinal disorders) | 2 (3)
Gastritis (Gastrointestinal disorders) | 1 (1)
Gastrointestinal disorders - Other, specify: Gastritis, reflux esophagitis, CMV postitve (Renal and urinary disorders) | 1 (1)
Hematuria (Hepatobiliary disorders) | 1 (1)
Hepatobiliary disorders - Other, specify: VOD (Respiratory, thoracic and mediastinal disorders) | 3 (3)
Hypoxia (Infections and infestations) | 1 (2)
Infections and infestations - Other, specify: CMV viremia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Klebsiella pneumoniae bacteremia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: RSV pneumonia (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Rotavirus gastroenteritis (Infections and infestations) | 1 (1)
Infections and infestations - Other, specify: Staphylococcus Epidermidis bacteremia (General disorders) | 1 (1)
Irritability (Infections and infestations) | 1 (1)
Lung infection (General disorders) | 1 (1)
Multi-organ failure (Musculoskeletal and connective tissue disorders) | 2 (3)
Musculoskeletal and connective tissue disorder - Other, specify: Cephalhematoma (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Pulmonary hypertension (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 4 (4)
Respiratory, thoracic and mediastinal disorders - Other, specify: Acute pulmonary hemorrhage (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: Bronchitis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: Chronic lung disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory, thoracic and mediastinal disorders - Other, specify: Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 2 (2)
Respiratory,thoracic and mediastinal disorders-Other:Abnormal CT chest;rulled out fungal disease (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory,thoracic and mediastinal disorders-Other:Bilateral pneumonia with pleural effusion (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Respiratory,thoracic and mediastinal disorders-Other:Respiratory distress secondary to fluid overloa (Nervous system disorders) | 1 (1) — Respiratory distress secondary to fluid overload
Seizure (Infections and infestations) | 2 (2)
Sepsis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Stridor (Infections and infestations) | 1 (1)
Upper respiratory infection (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify: Veno-occlusive disease (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Umbilical Cord Blood Transplant Treatment Plan (N=40)
Aspartate aminotransferase increased (Investigations) | 2 (3)
Bicarbonate, serum-low (Investigations) | 1 (1)
Blood bilirubin increased (Infections and infestations) | 4 (4)
Calcium, serum-low (hypocalcemia) (Investigations) | 1 (1)
Catheter related infection (Gastrointestinal disorders) | 6 (7)
Creatinine increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Diarrhea (Metabolism and nutrition disorders) | 2 (5)
Dyspnea (Metabolism and nutrition disorders) | 1 (1)
Fibrinogen (Vascular disorders) | 1 (1)
Hematuria (Metabolism and nutrition disorders) | 1 (1)
Hypermagnesemia (Metabolism and nutrition disorders) | 1 (1)
Hypernatremia (Metabolism and nutrition disorders) | 2 (5)
Hypertension (Metabolism and nutrition disorders) | 3 (4)
Hypertriglyceridemia (Metabolism and nutrition disorders) | 2 (5)
Hypoalbuminemia (Investigations) | 1 (1)
Hypocalcemia (Metabolism and nutrition disorders) | 7 (9)
Hyponatremia (Gastrointestinal disorders) | 4 (5)
Hypophosphatemia (Gastrointestinal disorders) | 2 (3)
INR (International Normalized Ratio of prothrombin time) (General disorders) | 1 (1)
Lipase increased (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Metabolism and nutrition disorders - Other, specify: Diabetic ketoacidosis (Respiratory, thoracic and mediastinal disorders) | 1 (1)
Mucositis oral (Skin and subcutaneous tissue disorders) | 1 (1)
Nausea (Nervous system disorders) | 1 (1)
PTT (Partial Thromboplastin Time) (Vascular disorders) | 1 (1)
Pain (Vascular disorders) | 1 (1)
Pharyngeal mucositis (Vascular disorders) | 1 (1)
Pulmonary edema (Vascular disorders) | 1 (1)
Rash maculo-papular (Vascular disorders) | 1 (1)
Seizure (Vascular disorders) | 3 (3)
Urinary tract infection (Vascular disorders) | 1 (1)
Vascular disorders - Other, specify: Thrombosis of left femoral vein (Vascular disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2021-06-01): https://cdn.clinicaltrials.gov/large-docs/46/NCT00950846/Prot_SAP_001.pdf
  • Informed Consent Form (2018-09-04): https://cdn.clinicaltrials.gov/large-docs/46/NCT00950846/ICF_000.pdf